CLINICAL TRIAL: NCT01157143
Title: Phase I, Double Blind, Parallel-Group, Multi-center, Gene Expression (Synthesis of FGF-1 mRNA) and Tolerability Study of Increasing Single Dose of NV1FGF Administered by Intra-Muscular Injection in Subjects With Severe Peripheral Artery Occlusive Disease (PAOD) Planned to Undergo Amputation Above the Ankle
Brief Title: Gene Expression and Tolerability Study of NV1FGF in Patients With Peripheral Artery Occlusive Disease Planned to Undergo Major Amputation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: International Clinical Development Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TED10105; PM105 (Other: Gencell)
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NV1FGF 500 μg (Experimental): 8 intramuscular injections for a total of 500 μg administered in one single administration 3 to 8 days before major amputation
  Interventions: Drug: XRP0038 (NV1FGF)
- NV1FGF 2000 μg (Experimental): 8 intramuscular injections for a total of 2000 μg administered in one single administration 3 to 8 days before major amputation
  Interventions: Drug: XRP0038 (NV1FGF)
- NV1FGF 4000 μg (Experimental): 8 intramuscular injections for a total of 4000 μg administered in one single administration 3 to 8 days before major amputation
  Interventions: Drug: XRP0038 (NV1FGF)

INTERVENTIONS:
Drug: XRP0038 (NV1FGF) — Pharmaceutical form : solution
  Route of administration : intramuscular

SUMMARY:
The primary objective is to evaluate the transgene expression (synthesis of FGF-1 mRNA) in injected tissue, at injection site, after Intra Muscular (IM) administration of increasing single doses of NV1FGF.

Secondary objectives :

* To evaluate the safety and tolerability of IM administration of increasing single doses of NV1FGF
* To evaluate the transgene expression (FGF-1 protein) in injected tissues (injection site and remote site)
* To evaluate the presence of FGF-1 receptors in injected tissues (injection site and remote site)
* To evaluate the NV1FGF biodistribution in injected tissues (injection site and remote site), in multiple organs/tissues when appropriate, and plasma
* To evaluate the transgene expression (synthesis of FGF-1 mRNA) in injected tissue at remote site
* To collect data from plasma NV1FGF pharmacokinetics
* To evaluate healing of the amputation site

DETAILED DESCRIPTION:
Screening of 1 to 4 weeks before study drug administration; Single study drug administration 3 to 8 days before planned amputation; 6 months of follow up

ELIGIBILITY:
Inclusion Criteria:

* Subjects with prior decision for amputation above the ankle because of severe PAOD
* Males or females above 18 years
* Females must be either:

  * Non pregnant, non lactating , having practicing a medically accepted method of birth control for more than 2 months prior screening visit;
  * or surgically sterilized (tubal ligation or hysterectomy)
  * or post menopausal for at least one year

Exclusion Criteria:

* Subjects with urgent need for amputation that cannot await until completion of the screening period (up to 4 weeks), added to the minimum required 48 hours between study test medication administration and tissue sample collection
* Previous or current history of malignant disease (subjects with successful tumor resection more than 5 years -without any recurrence- prior to study start could be enrolled)
* Abnormal Chest X-ray or mammography with suspicion of malignant disease
* Positive stool hemoccult (except in case of hemorrhoids or any other identified cause with no malignancy origin)
* Men with positive Prostate Specific Antigen (PSA) (above 2.5 ng/ml in subjects < 50 years and above 5 ng/ml in subjects above 50 years)
* Females with Papanicolaou smear of Class IV or Class V characterization
* Serious concomitant medical conditions not adequately controlled
* Alcohol or drug abuse
* Active proliferate retinopathy defined by the presence of new vessel formation and scarring
* Participation in clinical trials of non-approved experimental agents within four weeks before study entry;
* Positive serology for HIV1 or 2
* Creatinine above 2.0 mg/dl (176 µmol/l), unless the subject is on hemodialysis / peritoneal dialysis and diagnosed with complete and irreversible renal failure or end-stage renal disease (ESRD)
* Subjects who had a stroke or a neurological deficit presumably due to a stroke, within 3 months prior to study treatment (Amendment #1)
* Alpha-fetoprotein (AFP) in serum > 15 µg/l, unless liver ultrasound ruled out any malignant disease
* Positive serology for hepatitis B or C, unless liver ultrasound ruled out any malignant disease.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2002-01; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Detection of FGF-1 mRNA (by real-time RT-PCR) in injected tissues at injection site | 3 to 8 days after amputation

SECONDARY OUTCOMES:
Detection of FGF-1 protein (by immunohistochemistry) in injected tissues (injection and remote site) | 3 to 8 days after amputation
Detection of FGF-1 mRNA (by real-time RT-PCR) in injected tissues at remote site | 3 to 8 days after amputation
Detection of FGF-1 receptor (by immunohistochemistry) in injected tissues (injection and remote site) | 3 to 8 days after amputation
Detection of NV1FGF (by real-time PCR) in injected tissues (injection and remote site), in multiple organs/tissues when appropriate, and in plasma | 2 months
Evaluation of healing of the amputation site | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: International Clinical Development Clinical Study Director, Study Director — Sanofi
Locations (2):
- Minneapolis, Minnesota, United States
- Bern, Switzerland

REFERENCES:
- [Derived] Niebuhr A, Henry T, Goldman J, Baumgartner I, van Belle E, Gerss J, Hirsch AT, Nikol S. Long-term safety of intramuscular gene transfer of non-viral FGF1 for peripheral artery disease. Gene Ther. 2012 Mar;19(3):264-70. doi: 10.1038/gt.2011.85. Epub 2011 Jun 30. PMID 21716303